CLINICAL TRIAL: NCT00005062
Title: A Phase III Trial Comparing High Versus Standard Dose of Prophylactic Cranial Irradiation (PCI) in Limited Small Cell Lung Cancer Complete Responders
Brief Title: Radiation Therapy in Patients With Limited-Stage Small Cell Lung Cancer in Complete Remission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067664; FRE-IGR-PCI-99; EU-99051; FRE-IFCT-99.01; FRE-IGR-PCI99-EULINT1; EORTC-22003; EORTC-08004
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells and prevent the spread of cancer to the brain. It is not yet known if standard-dose radiation therapy is more effective than high-dose radiation therapy in preventing the spread of limited-stage small cell lung cancer cells to the brain.

PURPOSE: This randomized phase III trial is comparing two different regimens of radiation therapy to see how well they work in treating patients with limited-stage small cell lung cancer in complete remission.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare high-dose versus standard-dose prophylactic cranial radiotherapy in terms of the incidence of brain metastases and overall and disease free survival at 2 years in patients with limited stage small cell lung cancer in complete remission.
* Evaluate the quality of life and late sequelae in this patient population treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, age (60 and under vs over 60), and interval between the start of induction therapy and date of randomization (90 days or less vs 91-180 days vs more than 180 days). Patients are randomized into one of two treatment arms according to the prophylactic cranial radiotherapy dose.

* Arm I: Patients receive standard-dose prophylactic cranial radiotherapy (10 fractions/12 days).
* Arm II: Patients receive high-dose prophylactic cranial radiotherapy administered over 16 or 24 days based on the choice of their treatment center.

  * 18 fractions/24 days (conventional radiotherapy) OR
  * 24 fractions/16 days (accelerated hyperfractionated radiotherapy) Patients with isolated brain failure may undergo further radiotherapy.

Quality of life is assessed prior to randomization, at 6 months, at 1 year, and then annually thereafter.

Patients are followed at least every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 700 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven limited stage small cell lung cancer
* Complete response to induction therapy (at least on chest x-ray)
* Normal brain CT scan or MRI less than 1 month prior to study
* No metastases (including ipsilateral lung metastases and malignant pleural effusion)

PATIENT CHARACTERISTICS:

Age:

* 70 and under

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No prior cerebrovascular disease

Other:

* No epilepsy requiring permanent oral medication
* No other prior malignancy except skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No concurrent chemotherapy

Endocrine therapy:

* Concurrent steroids allowed

Radiotherapy:

* Concurrent thoracic radiotherapy allowed

Surgery:

* Not specified

Other

* No other concurrent antitumoral agent

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Incidence of brain metastases 2 years after randomization

SECONDARY OUTCOMES:
Overall survival and disease-free survival 2 years after randomization
Quality of life as assessed by Quality of Life Questionnaire (QLQ)-C30/BN20 before randomization, at 6 and 12 months, and annually thereafter
Treatment late sequelae as assessed by Late Effect of Normal Tissue - Subjective Objective Management Analytic scale, brain CT scan, or MRI before randomization and then annually thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Le Pechoux, MD — Gustave Roussy, Cancer Campus, Grand Paris; Suresh Senan — Free University Medical Center
Locations (93):
- M.D. Anderson Cancer Center at University of Texas, Houston, Texas, United States
- Australia (2):
  - Cancer Therapy Centre at Campbelltown Hospital, Campbelltown, New South Wales
  - Radiation Oncology Victoria, East Melbourne, Victoria
- Belgium (6):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Universiteit Gent, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
  - Clinique Saint-Joseph, Liège
  - Clinique Sainte Elisabeth, Namur
- Instituto Nacional de Cancer, Copacabana, Rio de Janeiro, Brazil
- Chile (2):
  - Instituto de Radiomedicina, Santiago
  - Clinica Renaca - Gocchi, Viña del Mar
- Rui Jin Hospital, Shanghai, China
- Hospital Militar Central, Bogotá, Colombia
- Bank Of Cyprus Oncology Centre, Nicosia, Cyprus
- Czechia (2):
  - Masaryk Memorial Cancer Institute, Brno
  - First Medical Clinic of Charles University Hospital, Prague
- France (33):
  - Clinique De Rochebelle, Alès
  - Centre de Traitement Hautes - Energies, Amiens
  - Centre Paul Papin, Angers
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - C.H.G. Beauvais, Beauvais
  - Polyclinique Bordeaux Nord Aquitaine, Boucher
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Radiotherapie, Compiègne
  - Centre Hospitalier Sud Francilien - Site Corbeil, Corbeil
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Hopital Intercommunal De Creteil, Créteil
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre De Radiotherapie Charlebourg, La Garenne-Colombes
  - Centre Guillaume Le Conquerant, Le Havre
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - C.R.T.T., Meudon-la-Forêt
  - C.H. General De Montbelliard, Montbelliard
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Institut Curie - Section Medicale, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Centre Frederic Joliot, Rouen
  - Centre du Rouget, Sarcelles
  - Centre Hospitalier Prive Des Yvelines, Sartrouville
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Centre Medico-Chirurgical Foch, Suresnes
  - Hopital d'Instruction des Armes Sainte-Anne, Toulon
  - Centre d'Oncologie Saint-Yves, Vannes
  - Institut Gustave Roussy, Villejuif
- Universitaetsklinikum Essen, Essen, Germany
- Greece (5):
  - University Hospital of Heraklion, Heraklion, Crete
  - Evaggelismos Hospital, Athens
  - Sotiria Hospital Chest Diseases, Athens
  - Venizelion Gr., Heraklion
  - University of Patras Medical School, Rio Patras
- Israel (2):
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - Ospedale Bellaria, Bologna
  - Universita Degli Studi Di Pisa, Pisa
  - Ospedale Ostetrico Ginecologica Sant Anna, Turin
- Osaka National Hospital, Osaka, Japan
- Institute of Oncology at Vilnius University, Vilnius, Lithuania
- Netherlands (4):
  - Akademisch Ziekenhuis Vrije Universiteit - Medisch Centrum, Amsterdam
  - Arnhems Radiotherapeutisch Instituut, Arnhem
  - Nijmegen Cancer Center at Radboud University Medical Center, Nijmegen
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
- Institute of Radiotherapy and Oncology, Skopje, North Macedonia
- Poland (4):
  - Medical University of Gdansk, Gdansk
  - Institute of Oncology, Lodz
  - Regional Lung Diseases Hospital, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
- Hospital Santa Maria, Lisbon, Portugal
- Institutul Oncologic - Universitatea de Medicina, Cluj-Napoca, Romania
- Institute of Oncology and Radiology of Serbia, Belgrade, Serbia
- Groote Schuur Hospital, Cape Town, South Africa
- Samsung Medical Center, Seoul, South Korea
- Spain (2):
  - Hospital Virgen de la Arrixaca, El Palmar
  - Hospital Virgen de las Nieves, Granada
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Marmara University Hospital, Istanbul, Turkey (Türkiye)
- United Kingdom (12):
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - New Cross Hospital, Wolverhampton, England
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Nevill Hall Hospital, Gwent, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales
  - Velindre Cancer Center at Velinde Hospital, Cardiff
  - Cancer Research Centre at Weston Park Hospital, Sheffield

REFERENCES:
- [Background] Le Pechoux C, Dunant A, Senan S, Wolfson A, Quoix E, Faivre-Finn C, Ciuleanu T, Arriagada R, Jones R, Wanders R, Lerouge D, Laplanche A; Prophylactic Cranial Irradiation (PCI) Collaborative Group. Standard-dose versus higher-dose prophylactic cranial irradiation (PCI) in patients with limited-stage small-cell lung cancer in complete remission after chemotherapy and thoracic radiotherapy (PCI 99-01, EORTC 22003-08004, RTOG 0212, and IFCT 99-01): a randomised clinical trial. Lancet Oncol. 2009 May;10(5):467-74. doi: 10.1016/S1470-2045(09)70101-9. Epub 2009 Apr 20. PMID 19386548
- [Background] Pechoux CL, Hatton M, Kobierska A, et al.: Randomized trial of standard dose to a higher dose prophylactic cranial irradiation (PCI) in limited-stage small cell cancer (SCLC) complete responders (CR): primary endpoint analysis (PCI99-01, IFCT 99-01, EORTC 22003-08004, RTOG 0212). [Abstract] J Clin Oncol 26 (Suppl 15): A-LBA7514, 2008.
- [Result] Le Pechoux C, Laplanche A, Faivre-Finn C, Ciuleanu T, Wanders R, Lerouge D, Keus R, Hatton M, Videtic GM, Senan S, Wolfson A, Jones R, Arriagada R, Quoix E, Dunant A; Prophylactic Cranial Irradiation (PCI) Collaborative Group. Clinical neurological outcome and quality of life among patients with limited small-cell cancer treated with two different doses of prophylactic cranial irradiation in the intergroup phase III trial (PCI99-01, EORTC 22003-08004, RTOG 0212 and IFCT 99-01). Ann Oncol. 2011 May;22(5):1154-1163. doi: 10.1093/annonc/mdq576. Epub 2010 Dec 7. PMID 21139020